CLINICAL TRIAL: NCT02040298
Title: A Phase II Randomized, Double-Blind, Parallel-Group, Placebo Controlled Crossover Trial to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of Clemastine Fumarate as a Remyelinating Agent in Multiple Sclerosis
Brief Title: Assessment of Clemastine Fumarate as a Remyelinating Agent in Multiple Sclerosis
Acronym: ReBUILD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ReBUILD
Record Dates: First submitted 2014-01-10; First posted 2014-01-20 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Clemastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 months Clemastine, 2 months Placebo (Active Comparator): 4mg clemastine twice daily for first 3 months -- crossover -- equivalent quantity/frequency of placebo for last 2 months
  Interventions: Drug: Clemastine; Drug: Placebo
- 3 months Placebo , 2 months Clemastine (Active Comparator): Placebo for first 3 months -- crossover -- 4mg clemastine twice daily for last 2 months.
  Interventions: Drug: Clemastine; Drug: Placebo

INTERVENTIONS:
Drug: Clemastine — 4mg tablet twice daily
  Other Names: Clemastine Fumarate,; Tavist -1
Drug: Placebo — Placebo tablet twice daily

SUMMARY:
The main purpose of this study is to assess clemastine as a remyelinating agent in patients with relapsing forms of multiple sclerosis. The study will also evaluate the tolerability of clemastine, originally approved as first-generation antihistamine, in patients with multiple sclerosis. Study procedures will include assessments for evidence of remyelination in the anterior visual pathway and in the brain using electrophysiologic techniques and magnetic resonance imaging. The study will also assess the robustness and stability of this clinical effect in patients taking clemastine for up to 3 months. Patients in this study can remain on their standard disease modifying treatment during the course of the study. However, patients cannot participate in any other investigational new drug research study concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting Multiple Sclerosis by 2010 Revised McDonald Criteria
* Age 18-60.
* Latency delay > 125 milliseconds on baseline full-field transient pattern reversal visual evoked potential (VEP) in at least one eye (electrophysiological evidence of demyelination)
* Retinal nerve fiber layer (RNFL) > 70 microns on Spectralis Domain Optical Coherence Topography (SD-OCT) in the same eye meeting criteria for latency delay (sufficient axons)
* No optic neuritis in prior 6 months
* Stable immunomodulatory therapy - no switch or planned switch in > 6 months and no change in doses in 30 days prior to screening
* Use of appropriate contraception during period of trial (females of child bearing potential)
* Understand and sign informed consent.
* Expanded disability status scale (EDSS) 0-6.0 (inclusive)

Exclusion Criteria:

* Major ophthalmologic disease / Concomitant ophthalmologic disorders (e.g. diabetes, macular degeneration, glaucoma, severe myopia , etc).
* Myopia > -7 Diopters (Severe myopia)
* History of significant cardiac conduction block
* History of cancer
* Known optic neuritis in involved eye > 5 years ago OR disease duration > 15 years
* Suicidal ideation or behaviour in 6 months prior to screening
* Pregnancy, breastfeeding, or planning to become pregnant.
* Involved with other study protocol simultaneously without prior approval. 9. Concomitant use of Dalfampridine (4AP or diamino4AP) or any other formulation of 4AP or diamino4AP.
* Concomitant use of any other putative remyelinating therapy as determined by investigator.
* Treatment with corticosteroids within 30 days prior to screening
* Prior treatment with total lymphoid irradiation, T cell or T cell receptor vaccination
* Prior treatment with alemtuzumab, mitoxantrone, or cyclophosphamide
* Serum creatinine > 1.5 mg/dL; aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase > 2 times the upper limit of normal
* History of drug or alcohol abuse within the past year
* Untreated vitamin B12 deficiency (as determined by B12 serological assessments and metabolites including methylmalonic acid (MMA) and homocysteine) or untreated hypothyroidism
* Clinically significant cardiac, metabolic, hematologic, hepatic, immunologic, urologic, endocrinologic, neurologic, pulmonary, psychiatric, dermatologic, psychiatric allergic, renal or other major diseases that in the PI's judgment may affect interpretation of study results or patient safety.
* History of or presence of clinically significant medical illness or laboratory abnormality that, in the opinion of the investigator would preclude participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari J. Green, MD, MCR, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Multiple Sclerosis Center, San Francisco, California, United States

REFERENCES:
- [Background] Fischer JS, LaRocca NG, Miller DM, Ritvo PG, Andrews H, Paty D. Recent developments in the assessment of quality of life in multiple sclerosis (MS). Mult Scler. 1999 Aug;5(4):251-9. doi: 10.1177/135245859900500410. PMID 10467384
- [Result] Green AJ, Gelfand JM, Cree BA, Bevan C, Boscardin WJ, Mei F, Inman J, Arnow S, Devereux M, Abounasr A, Nobuta H, Zhu A, Friessen M, Gerona R, von Budingen HC, Henry RG, Hauser SL, Chan JR. Clemastine fumarate as a remyelinating therapy for multiple sclerosis (ReBUILD): a randomised, controlled, double-blind, crossover trial. Lancet. 2017 Dec 2;390(10111):2481-2489. doi: 10.1016/S0140-6736(17)32346-2. Epub 2017 Oct 10. PMID 29029896
- [Derived] Abdelhak A, Cordano C, Boscardin WJ, Caverzasi E, Kuhle J, Chan B, Gelfand JM, Yiu HH, Oertel FC, Beaudry-Richard A, Condor Montes S, Oksenberg JR, Lario Lago A, Boxer A, Rojas-Martinez JC, Elahi FM, Chan JR, Green AJ. Plasma neurofilament light chain levels suggest neuroaxonal stability following therapeutic remyelination in people with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2022 Jun 16:jnnp-2022-329221. doi: 10.1136/jnnp-2022-329221. Online ahead of print. PMID 35710320
- See also: ReBUILD trial description University of California, San Francisco Multiple Sclerosis Center — http://multiplesclerosis.ucsf.edu/research/rebuild

RESULTS

PARTICIPANT FLOW:
Groups:
- Clemastine First, Then Placebo: Participants first received Clemastine 4mg twice daily for 3 months. Then they received Placebo (matching Clemastine 4mg) twice daily for 2 months.
- Placebo First, Then Clemastine: Participants first received Placebo (matching Clemastine 4mg) twice daily for 3 months. Then they received Clemastine 4mg twice daily for 2 months.
Period: First Intervention (3 Months)
Arm/Group | Clemastine First, Then Placebo | Placebo First, Then Clemastine
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention (2 Months)
Arm/Group | Clemastine First, Then Placebo | Placebo First, Then Clemastine
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clemastine First, Then Placebo: Participants first received Clemastine 4mg tablet twice daily for 3 months, then they received Placebo (matching Clemastine 4mg) for 2 months.
- Placebo First, Then Clemastine: Participants first received Placebo (matching Clemastine 4mg) tablet twice daily for 3 months, then they received Clemastine 4mg twice daily for 2 months.
- Total: Total of all reporting groups
Arm/Group | Clemastine First, Then Placebo | Placebo First, Then Clemastine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (10.8) | 40.0 (10.1) | 40.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 6 | 12 | 18
Disease duration [Mean (Standard Deviation); unit: years] | 5.7 (6.5) | 4.4 (3.6) | 5.1 (5.2)
EDSS [Mean (Standard Deviation); unit: units on a scale] — Expanded Disability Status Scale (EDSS) is an ordinal scale for assessing neurological impairment of MS based on a neurological examination. It consists of scores in each of seven functional systems (FS) and an ambulation score that are then combined to determine the EDSS [ranging from 0 (normal) to 10 (death due to MS)].
  units on a scale | 2.2 (1.0) | 2.1 (1.2) | 2.2 (1.1)
History of optic neuritis [Count of Participants; unit: Participants] | 15 | 13 | 28
Time since optic neuritis [Mean (Standard Deviation); unit: years] | 3.7 (3.4) | 4.9 (4.6) | 4.3 (4.0)
VEP P100 latency [Mean (Standard Deviation); unit: milliseconds] — Visual Evoked Potential (VEP); prominent positive deflection (P100)
  milliseconds | 128.6 (11.6) | 126.8 (9.4) | 127.7 (10.5)
OCT Retinal Nerve Fiber Layer (RNFL) [Mean (Standard Deviation); unit: µm] — Optical Coherence Tomography (OCT) Retinal Nerve Fiber Layer (RNFL)
  µm | 90.2 (12.0) | 85.1 (7.9) | 86.7 (10.4)
OCT Macular volume [Mean (Standard Deviation); unit: mm^3] | 3.05 (0.14) | 3.01 (0.11) | 3.03 (0.13)
LCLA [Mean (Standard Deviation); unit: Number of letters read correctly] — Low Contrast Letter Acuity (LCLA) is scored from 0-70. Higher scores are better.
  Number of letters read correctly | 24.0 (8.4) | 21.6 (10.7) | 22.8 (9.6)
SDMT [Mean (Standard Deviation); unit: number of correct substitutions] — Symbol Digit Modalities Test (SDMT) is scored 0-110. Higher scores are better.
  number of correct substitutions | 51.8 (10.2) | 50.0 (11.1) | 50.9 (10.6)
MAF [Mean (Standard Deviation); unit: units on a scale] | 17.82 (12.39) | 20.43 (10.88) | 19.13 (11.62)
6-min walk [Mean (Standard Deviation); unit: feet] | 1742.40 (288.14) | 1741.76 (260.08) | 1742.08 (271.66)
25-foot walk [Mean (Standard Deviation); unit: seconds] | 3.81 (0.67) | 4.10 (1.01) | 3.96 (0.86)
Myelin water fraction [Mean (Standard Deviation); unit: ratio] | 67.55 (11.85) | 65.70 (12.98) | 66.62 (12.33)
MTR 25 [Mean (Standard Deviation); unit: ratio]
  Brain | 0.39 (0.05) | 0.38 (0.03) | 0.39 (0.04)
  White matter | 0.54 (0.02) | 0.54 (0.02) | 0.54 (0.02)
FA white matter [Mean (Standard Deviation); unit: ratio] | 0.24 (0.02) | 0.24 (0.01) | 0.24 (0.01)

OUTCOME MEASURES:

1. Primary Outcome: Full Field Visual Evoked Potential (VEP)
Description: The primary objective is to evaluate the efficacy of Clemastine relative to placebo for reducing P100 latencies on full field transient pattern reversal visual evoked potentials.Visual evoked potentials (VEP) are used primarily to measure the functional integrity of the visual pathways from the retina to the visual cortex of the brain. VEP latencies were collected at Baseline, Month 1, Month 3, and Month 5.
Time Frame: Treatment start to treatment end, up to 3 months.
Population: The data for 7 eyes did not meet criteria for inclusion in analysis (i.e., absent or unidentifiable waveforms.).
Measure: Mean (Standard Deviation); unit: ms
Units Other Than Participants: eyes
Groups:
- Clemastine: Participants who received clemastine 4mg twice daily in either the first 3 months or the last 2 months of the study
- Placebo: Participants who received Placebo tablet (matching clemastine 4mg) twice daily in either the first 3 months or last 2 months of the study.
Arm/Group | Clemastine | Placebo
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 93 | 93
ms
  VEP at baseline | 124.8 (11.5) | 126.4 (10.9)
  VEP change from baseline | -2.86 (6.85) | -1.50 (3.86)

2. Secondary Outcome: Tolerability of Clemastine in Multiple Sclerosis (MS) Patients
Description: Will demonstrate the tolerability of Clemastine in this population. This will include special focus with regards to fatigue as this is a major symptom for patients suffering from multiple sclerosis.This will be assessed by administering a fatigue questionnaire called the Multidimensional Assessment of Fatigue (MAF) at all four visits throughout the study. MAF scale range is 0-50. Lower scores indicate lower levels of fatigue and higher scores indicate higher levels of fatigue.
Time Frame: Treatment start to treatment end, up to 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Clemastine: Participants who received clemastine 4mg tablet twice a day either the first 3 months or last 2 months of the study.
- Placebo: Participants who received Placebo (matching clemastine 4mg) twice a day in either the first 3 months or last 2 months of the study.
Arm/Group | Clemastine | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  MAF at baseline | 21.0 (10.9) | 18.8 (12.2)
  MAF change from baseline | 1.9 (6.8) | -0.4 (6.9)

3. Secondary Outcome: Myelin Water Fraction (MWF) and Magnetization Transfer Ratios (MTR)
Description: To evaluate the efficacy of Clemastine relative to placebo in increasing magnetization transfer ratios derived from magnetic resonance imaging (MRI) of the brain during the period of exposure to active treatment.
  To evaluate the efficacy of Clemastine relative to placebo at reducing radial diffusivity derived from diffusion tensor imaging as assessed by magnetic resonance imaging (MRI) during the period of exposure to active medication.
Time Frame: Treatment start to treatment end, up to 3 months.
Population: MRI done at baseline, month 3, month 5
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Clemastine: Participants who received Clemastine 4mg tablet twice daily in either the first 3 months or the last 2 months of the study.
- Placebo: Participants who received Placebo (matching clemastine 4mg tablet) in either the first 3 months or the last 2 months of the study.
Arm/Group | Clemastine | Placebo
Number analyzed (Participants) | 50 | 50
Ratio
  MTR 25: full brain at baseline | 0,380 (0.040) | 0.379 (0.041)
  MTR: white matter at baseline | 0.533 (0.018) | 0.533 (0.021)
  MWF 50 at baseline | 66.38 (13.06) | 66.12 (12.69)
  MTR 25: full brain change from baseline | -0.008 (0.016) | -0.009 (0.018)
  MTR: white matter change from baseline | -0.004 (0.021) | -0.004 (0.018)
  MWF 50 change from baseline | 0.23 (13.20) | -0.55 (10.78)

4. Secondary Outcome: Expanded Disability Status Scale (EDSS) Score
Description: To evaluate the efficacy of Clemastine relative to placebo in reducing the EDSS score at 90 days compared to placebo (Group A) & at 150 days compared to day 90 (Group B). EDSS is an ordinal scale for assessing neurological impairment of MS based on a neurological examination. It consists of scores in each of seven functional systems (FS) & an ambulation score that are then combined to determine the EDSS [ranging from 0 (normal) to 10 (death due to MS)]. The FSs are the Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, & Cerebral functions. FSs & EDSS steps assessed in a standardized manner. EDSS is a widely used &accepted instrument to evaluate disability status at a given time & longitudinally, to assess disability progression in clinical studies in MS.
Time Frame: Start of treatment to end of treatment, up to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Clemastine: Participants who received Clemastine 4mg tablet twice daily in either the first 3 months or last 2 months of the study.
- Placebo: Participants who received Placebo (matching Clemastine 4mg) in either the first 3 months or last 2 months of the study.
Arm/Group | Clemastine | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  EDSS at baseline | 2.06 (1.21) | 2.14 (1.15)
  EDSS change from baseline | -0.09 (0.87) | -0.03 (0.69)

5. Other Pre Specified Outcome: Serum Creatinine Level
Description: Blood sample will be collected at each visit to evaluate health status...
Time Frame: Baseline, 1 month, 3 month, 5 month
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Serum Triglyceride Level
Description: Blood sample will be collected at each visit to evaluate health status.
Time Frame: Baseline, 1 month, 3 month, 5 month
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Vitamin B-12 Level
Description: Blood sample will be collected at each visit to evaluate health status.
Time Frame: Baseline, 1 month, 3 month, 5 month
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Human Chorionic Gonadotropin (hCG) Level in Female Patients of Childbearing Potential
Description: Blood and urine sample will be collected to assess pregnancy status of all female participants of child bearing potential.
Time Frame: Baseline, 1 month, 3 month, 5 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 months.
Groups:
- Clemastine: Participants received Clemastine 4mg twice daily for either 3 months or 2 months.
- Placebo: Participants received Placebo (matching Clemastine 4mg) for either 3 months or 2 months.
Arm/Group | Clemastine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 10/50 | 15/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clemastine (N=50) | Placebo (N=50)
Increased trigylcerides (Investigations) | 10 | 14
Severe fatigue (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes